CLINICAL TRIAL: NCT00238563
Title: Post-Operative Sub-Tenon Kenalog in Glaucoma Filtering Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not secured
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 7/8/05-21
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone injection, sub-tenon

SUMMARY:
Determine efficacy of sub tenon kenalog injections for post-operative management of trabeculectomy procedures.

DETAILED DESCRIPTION:
Postoperative sub-Tenon Triamcinolone Acetonide in glaucoma filtering surgery

Objectives: Trabeculectomy is a surgical procedure designed to reduce internal eye pressure by draining fluid from within the eye to the sub-conjunctival (superficial eye lining) space. Scar formation from conjunctival and Tenon's capsule fibroblast proliferation represents the most common cause of failure of trabeculectomies. A number of drugs have been use to prevent failure of trabeculectomies from the scarring process including intraoperative mitomycin C (MMC) and preoperative Triamcinalone Acetonide (TA). Over the past several years, intraoperative MMC has become a preferred method of preventing scar formation. This study looks to determine in a prospective, double-blind, randomized method the long-term efficacy and safety of MMC with postoperative TA compared to the standard practice of intraoperative MMC with postoperative prednisolone acetate drops in preventing scar related failures of trabeculectomies.

ELIGIBILITY:
Inclusion Criteria:Trabeculectomy surgery patient, age 18 or older - Exclusion Criteria:Pregnant, nursing, age less than 18, known allergy to medication being studied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure

SECONDARY OUTCOMES:
visual field progression, need for further surgery or medications

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Santa Clara valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California